CLINICAL TRIAL: NCT00902967
Title: A Randomized Double Blind Study Of The Evaluation Of The Potential Analgesic And Anti-Inflammatory Effects Of Atorvastatin In Patients Undergoing Abdominal Surgery
Brief Title: Study To Check The Analgesic And Anti-Inflammatory Effects Of Atorvastatin In Patients Undergoing Abdominal Surgery
Acronym: A4S
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: B. J. Medical College, Pune (Other)
Responsible Party: Dr Bharati Daswani, Assosiate Proffessor, Department of Pharmacology, B. J. medical College & Sassoon General Hospitals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASU 1
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Abdominal Surgery
Keywords: Postoperative pain; atorvastatin; analgesic; antiinflammatory
MeSH Terms: conditions — Pain, Postoperative | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Tablet Atorvastatin 10 mg once daily for 5 weeks (1 week before operation till 2 weeks after the operation)
  Interventions: Drug: Atorvastatin
- 2 (Placebo Comparator): Placebo tablets of similar shape and color given at night time dosing
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 10 mg, once a day dosing at night after meals
  Arms: 1
Drug: Placebo — Placebo tablets of similar shape size and color given once a day at night time after meals
  Arms: 2

SUMMARY:
The study is planned to check the analgesic and anti-inflammatory properties of Atorvastatin in patients who will be undergoing abdominal surgery under spinal anesthesia. The investigators intend to monitor the analgesic requirements, the rate of wound healing and the inflammatory markers in this trial.

DETAILED DESCRIPTION:
Study type: Double Blind Placebo Controlled

Method of Randomization: Computer Generated Table

No. of patients to be recruited: 40

Accept Healthy Volunteers: No

Drugs to be administered: Atorvastatin to 20 patients and placebo to 20 patients

Mode of drug administration: Oral

Duration of Study: 3 weeks

Patients who attend the Surgical O.P.D and the Obstetrics and Gynaecology O.P.D and are diagnosed with any condition that requires elective abdominal surgery under spinal anaesthesia will be chosen for screening. Patients undergoing day care surgery with spinal anaesthesia and an abdominal incision will also be included for screening.

Two weeks before the decided date of surgery the patients will be called for screening. The patients will first be screened for obesity, risk factors for CVS diseases and blood will be withdrawn for estimation of serum lipid levels. Further risk assessment of these patients will be done according to the NCEP ATP III Guidelines (2004 Revision of NCEP Adult Treatment Panel III Guidelines). If the patient is under the moderate risk category and fits in the inclusion criteria he/she will be called the next week for starting atorvastatin/placebo.

Patients who are defined as dyslipidemic in the moderate risk category according to NCEP ATP III Guidelines i.e patients who would benefit from statin therapy will be given atorvastatin 10 mg or placebo started one week before their expected date of surgery. They will be explained the possible A.D.R of statin therapy. Informed consent form will be filled.

On the day of the surgery the patient will be explained the Visual Analouge Scale and the Wong Pain Scale. After the operation the patients will be started on S.O.S analgesic therapy. The protocol used will be the same as followed in the surgical wards. In case of severe pain opioids will be used. For other types of pain which can be tolerated by the patients Diclofenac Sodium will be used.

The patient will be monitored after the surgery for the total dose of analgesics required for the relief of pain. Further the time of first dose of analgesic required after operation will be noted. The patient will be monitored for pain at the incision site 2, 4, 6, 12, 24 hours after the operation using the visual analogue scale and the Wong Pain Scale. Later using the abovementioned scales the patient's pain will be monitored twice daily until the patient is discharged. The McGill Pain Questionnaire will be given to the patient on the first day and every day thereafter till the patient is discharged. After discharge the patient will followed up on the day of their suture removal and pain scores will be evaluated. The patient will be asked to come weekly till the end of the study period.

Blood will be withdrawn for the estimation of serum lipid levels, total leukocyte counts, C - reactive protein and TNF-α levels at baseline(i.e day of starting therapy), on the day of the surgery before the surgery and at the fourth postoperative day. All blood samples will be taken between 10A.M-12P.M Wound healing will be monitored on a daily basis until discharge and weekly thereafter. The attending surgeon will monitor the wound for discharge, swelling, etc. Additional signs of inflammation and infection like swelling, fever, erythema will also be monitored for.

The patients will be instructed to take atorvastatin or placebo once a day for three weeks (One week preoperative and two weeks postoperative). At the end of this period the patient will be asked to continue statins from outside. In the event that the patient is unable to afford the medication he will be weaned off the statin in a gradual manner.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 25-55 years
2. Patients who will be undergoing abdominal surgery under spinal anaesthesia
3. Patients who will undergo non-bowel abdominal surgery with an abdominal incision
4. Understands and agrees to comply with all study procedures including the daily treatments and follow-up visits
5. Able to understand and is voluntarily willing to sign an informed consent form for this study
6. Weight between 50 and 120 kg

Exclusion Criteria:

1. Bowel surgery or surgery under general anaesthesia
2. Any emergency operations
3. Surgery in patients in whom the chances of infection are very high. Example peritonitis, cystitis, appendical abscess, perforations, etc
4. Laparoscopic Surgery
5. Pregnant or nursing, or with the ability to become pregnant and not using an accepted form of birth control
6. Any active Cancer
7. Uncontrolled diabetes mellitis
8. Untreated hypertension
9. Psychotic disorder(s), dementia, mental retardation, or other organic mental disorders (subjects who are not mentally and physically able to personally consent for participation in this study are not eligible)
10. Any other (including acute) condition, which in the opinion of the investigator, is likely to cause non-compliance or significantly impact treatment outcomes
11. Sensitivity to the study drug or its components

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-12 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Pain as measured on Visual Analogue Scale | 2, 4, 6, 12, 24 hour post-operative and twice daily till discharge

SECONDARY OUTCOMES:
Pain measured on Wong Pain Scale | 2, 4, 6, 12, 24 hours post-operative and twice daily thereafter till discharge
Pain measured by the McGill Pain Questionnaire | Once daily till discharge
TNF Alpha Levels | baseline, on day of surgery, day 4 postoperative
Serum Lipid Levels | Before starting Atorvastatin and at end of study
C Reactive Protein Levels | baseline, on day of surgery, day 4 postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pharmacology, Sassoon General Hospitals, Pune, Maharashtra, India